CLINICAL TRIAL: NCT02007031
Title: Cardiovascular Responses to Cold Exposure in Hypertension
Brief Title: Cardiovascular Responses to Cold in Hypertension
Acronym: ColdHTN
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Finnish Institute of Occupational Health (Other); Verve Research, Oulu, Finland (Other)
Responsible Party: Principal Investigator, Tiina Ikäheimo, Postdoctoral researcher, University of Oulu
Other Study IDs: 24300771KYTEM
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
Keywords: Hypertension; Cold temperature; Blood pressure; Electrocardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypertensive subjects: Hypertensive subjects are exposed to brief cold exposure (-15 C for 15 min) mainly subjected to their facial region during which their cardiovascular responses are registered.
- Normotensive subjects: Normotensive subjects are exposed to brief cold exposure (-15 C for 15 min) mainly subjected to their facial region during which their cardiovascular responses are registered.

SUMMARY:
Wintertime is associated with increased morbidity and mortality and a majority is related to cardiovascular causes, such as myocardial infarctions, heart failures, and strokes. It is also known, that both acute and long-term cold exposure increase blood pressure and cardiac workload, and this may contribute to the observed excess morbidity and mortality during the cold season.

Although the effects of cold on blood pressure are known among healthy people, these responses among risk groups, such as hypertensive people, are not established. In addition, changes in cardiac electrical activity or autonomic regulation are largely unknown. The cardiovascular responses in the cold could be different among hypertensive people because of disturbances in the circulatory regulation or function, such as aortic stiffening and increased vasomotor tone of peripheral arteries due to endothelial dysfunction associated with the disease. To assess this, a controlled experiment employing a cold exposure similar to everyday winter circumstances in a subarctic climate was performed.

DETAILED DESCRIPTION:
Introduction.

Wintertime is associated with increased morbidity and mortality and a majority is related to cardiovascular causes, such as myocardial infarctions, heart failures, and strokes. It is also known, that both acute and long-term cold exposure increase blood pressure and cardiac workload, and this may contribute to the observed excess morbidity and mortality during cold season.

Although the effects of cold on blood pressure are established among healthy people, the effects among risk groups, such as hypertensive people, are not known. In addition to blood pressure, information on cardiac electrical activity or autonomic regulation are needed. Cardiovascular responses in the cold could be different among hypertensive people because of disturbances in autonomic nervous system and the circulatory regulation or function, such as aortic stiffening and increased vasomotor tone of peripheral arteries due to endothelial dysfunction associated with the disease. To assess this, a controlled experiment employing a cold exposure similar to everyday winter circumstances in a subarctic climate was performed in a climatic chamber.

Aims of the research.

The objective of the research was to assess how short-term cold exposure affects cardiovascular function of middle-aged untreated hypertensive and normotensive men. The hypotheses of the study were: a) cold exposure induces adverse changes in cardiovascular function, such as higher blood pressure and cardiac workload and b) hypertensive men demonstrate an aggravated response to cold exposure and the recovery of the cardiovascular system to baseline is delayed compared to normotensive subjects.

Material and Methods.

Study participants.

The study participants were chosen through a population-based recruitment and where a random sample of 1000 men (55-65 years old) living in Oulu, Finland was drawn from the Finnish Population Register. The subjects were screened by telephone interviews for eligibility for the study. Eligible attendees measured their blood pressure at home for a week according to the recommendations of the European Society of Hypertension. Based on these measurements they were classified either to hypertensive (systolic blood pressure ≥135 and/or diastolic blood pressure ≥85 mmHg) or normotensive (blood pressure <135/85mmHg).(16) The exclusion criteria was the presence of coronary heart or respiratory diseases, use of antihypertensive drugs for any indication, an average home BP ≥175/105 mm Hg, and failed home BP measurements. We aimed at recruiting a 2:1 ratio of hypertensive and normotensive subjects. The final study group consisted of 56 hypertensive and 35 normotensive middle-aged men.

Measurement protocol.

Before the measurements the participants filled a questionnaire with health and cold habituation related questions. The laboratory experiments began with a short familiarization to the measurement protocol and climatic chambers. Height, body composition, and physical fitness of the subjects were measured.

The participants were exposed for 15 min to temperature of -10°C and wind of 3m/s while protected from the cold with proper winter clothing, i.e. conditions similar to common habitual winter time cold exposure in subarctic countries. Participants were followed 15 min before (control measurements) and 20 min after (recovery) the exposure in a climatic chamber where the temperature was adjusted to +18°C and wind was set to <0.2m/s). The participants were standing with their arms supported during the measurements.Cardiovascular function was assessed by measuring brachial, central aortic, and continuous "beat to beat" blood pressure, as well as ECG measurements. The intensity of cold exposure was evaluated with skin temperature measurements (middle finger, back of the hand, shoulder blade, and cheek) and by assessing thermal perception for the whole body and face using subjective judgement scales.

The collected data was analyzed to assess the cold related changes in blood pressure (brachial and central aortic) and heart rate. ECG morphology and vector cardiographic parameters were computed from derived 12-lead ECG recordings at the Institute of Clinical Medicine at University of Oulu. Arrhythmias were detected automatically and confirmed with visual inspection by trained health care professional. To assess the regulation of circulation, continuous blood pressure signal and simultaneously recorded three lead ECG are applied to compute baroreflex sensitivity and heart rate variability at the Verve research center. In the data analyses responses to cold exposure will be evaluated and compared between hypertensive and normotensive subjects. In addition to the above mentioned topics combined risk factors for adverse changes in cardiovascular function during cold exposure will be evaluated, such as high arterial stiffness, altered ECG, and low heart rate variability. Based on this, a profile of a high risk patient will be defined and shared with physicians treating hypertensive patients to reduce adverse cold-related cardiac events.

Site of research and availability of equipment and services required for the research.

The laboratory measurements were implemented in the climatic chambers of Kastelli Research Center, Oulu, Finland. The data analyses and reporting are performed in facilities of Center for Environmental and Respiratory Health Research (University of Oulu). In addition, data analyses are performed in the Oulu University Hospital and at Verve department of Exercise and Cardiac rehabilitation.

Co-operation.

The Center for Environmental and Respiratory Health Research - Adjunct professor Tiina M Ikäheimo, Professor Jouni JK Jaakkola, Professor J Hassi, PhD A Rantala, MHSc H Hyrkäs; Department of Exercise and Medical Physiology, Verve, Oulu - Adjunct professor M Tulppo, Adjunct professor A Kiviniemi, Adjunct professor Arto Hautala; Institute of Occupational Health, Oulu - Professor H Rintamäki; Institute of Clinical Medicine, University of Oulu - Professor H Huikuri, PhD T Kenttä; Institute of Biomedicine, Department of Physiology and Biocenter of Oulu, University of Oulu - Professor KH Herzig; Institute of Health Sciences, University of Oulu - Professor S Keinänen-Kiukaanniemi, Professor R Antikainen, Professor M Mäntysaari; Department of Biology - Professor E Hohtola; Oulu University of Applied Sciences - Principal lecturer of Medical Engineering J Jauhiainen.

Ethical issues.

The study was approved by the ethics committee of Northern Ostrobothnia Hospital District (statement number 240/2010) and all participants were informed of the study and were requested for informed consent. They had also the possibility to terminate the study at any point. The data collected during the study is maintained unavailable from other than project personnel and protected with passwords. Data-analyses are performed without any personal identification (name, address etc.). The research applied a short cold exposure with well protected subjects and did not, therefore, cause any pain or harm to the participants.

Implications.

WHO has defined high blood pressure as the leading global risk for mortality in the world. Approximately half of the middle-aged men and one third of women have hypertension in Finland. On the other hand, with proper blood pressure control the risk of adverse cardiovascular events among hypertensive patients can be considerably reduced.

Wintertime and cold weather remarkably increase the risk of cardiovascular morbidity and mortality. There is an excess of ca. 2000-3000 deaths occurring in Finland during the winter and even half of them are for cardiovascular reasons. Both acute and and repeated exposures to cold increase blood pressure and may contribute to the higher wintertime cardiovascular morbidity and mortality. It has been suggested, that cold-related cardiovascular deaths could be prevented by proper protection from cold temperature.

The study will produce novel information of cardiovascular responses to short-term cold exposure among untreated hypertensive men. This knowledge will help health care personnel to advice hypertensive patients to protect themselves during habitual cold exposure, which could reduce the adverse cardiac events related to the cold weather. This knowledge is useful for medical doctors when considering medication for their patients. In addition, hypertensive people may need advice for their proper protection to reduce cold-related changes in cardiovascular function, such as blood pressure increases, and the related adverse cardiovascular events in cold climates.

ELIGIBILITY:
Inclusion Criteria:

* Measured BP (home measurements of one week) above 135/85 mmHg were selected to the group of hypertensive subjects.
* Those with BP below 135/85 mmHg were selected as controls.

Exclusion Criteria:

* Presence of coronary heart disease, respiratory diseases, and the use of antihypertensive drug treatment.
* an average home BP ≥175/105 mmHg, initiating antihypertensive drug treatment, failed home BP measurements, and having a respiratory infection within a week prior to the controlled measurements

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants were included according to a population based recruitment where a random sample of 1000 men (55-65 years old) living in Oulu, Finland was drawn from the Finnish Population Register. They were screened by telephone interviews for eligibility for the study. Eligible attendees measured their blood pressure home for a week according to the recommendations of the European Society of Hypertension and were classified either to hypertensive (systolic blood pressure ≥135 and/or diastolic blood pressure ≥85 mmHg) or normotensive (blood pressure <135/85mmHg). For the study we aimed at a 2:1 ratio of hypertensive and normotensive. The final study group consisted of 56 hypertensive and 35 normotensive middle-aged men.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure response of hypertensive and normotensive subjects to cold exposure | 2 hours (measured within the controlled experiment)
  The study assesses the blood pressure response of hypertensive and normotensive subjects to facial cooling. Blood pressure is measured before (warm, +18°C), during (cold, 15°C) and after (warm, +18°C) the employed cold exposure. The duration of each of these exposures are 30, 15 and 30 min.

SECONDARY OUTCOMES:
Cardiac autonomic regulation | 2 hours (measured within each controlled experiment), ECG recorded continuously
  ECG is recorded continuously during the controlled experiment (15 min warm 18 C, 15 min cold exposure -15 C and 20 min 18 C) from where cardiac electrical function, as well as autonomic nervous system regulation is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Ikäheimo, Ph.D., Principal Investigator — University of Oulu; Jouni JK Jaakkola, MD, Ph.D., Principal Investigator — University of Oulu
Locations (2):
- Finland (2):
  - University of Oulu, Oulu
  - Finnish Institute of Occupational Health, Oulu

REFERENCES:
- [Background] Ikaheimo TM, Lehtinen T, Antikainen R, Jokelainen J, Nayha S, Hassi J, Keinanen-Kiukaanniemi S, Laatikainen T, Jousilahti P, Jaakkola JJ. Cold-related cardiorespiratory symptoms among subjects with and without hypertension: the National FINRISK Study 2002. Eur J Public Health. 2014 Apr;24(2):237-43. doi: 10.1093/eurpub/ckt078. Epub 2013 Jun 22. PMID 23794677
- [Background] Edwards DG, Gauthier AL, Hayman MA, Lang JT, Kenefick RW. Acute effects of cold exposure on central aortic wave reflection. J Appl Physiol (1985). 2006 Apr;100(4):1210-4. doi: 10.1152/japplphysiol.01154.2005. Epub 2005 Oct 13. PMID 16223975
- [Background] Modesti PA, Morabito M, Massetti L, Rapi S, Orlandini S, Mancia G, Gensini GF, Parati G. Seasonal blood pressure changes: an independent relationship with temperature and daylight hours. Hypertension. 2013 Apr;61(4):908-14. doi: 10.1161/HYPERTENSIONAHA.111.00315. Epub 2013 Feb 4. PMID 23381792
- [Background] Barnett AG, Sans S, Salomaa V, Kuulasmaa K, Dobson AJ; WHO MONICA Project. The effect of temperature on systolic blood pressure. Blood Press Monit. 2007 Jun;12(3):195-203. doi: 10.1097/MBP.0b013e3280b083f4. PMID 17496471
- [Background] Barnett AG, Dobson AJ, McElduff P, Salomaa V, Kuulasmaa K, Sans S; WHO MONICA Project. Cold periods and coronary events: an analysis of populations worldwide. J Epidemiol Community Health. 2005 Jul;59(7):551-7. doi: 10.1136/jech.2004.028514. PMID 15965137
- [Background] Parati G, Stergiou GS, Asmar R, Bilo G, de Leeuw P, Imai Y, Kario K, Lurbe E, Manolis A, Mengden T, O'Brien E, Ohkubo T, Padfield P, Palatini P, Pickering TG, Redon J, Revera M, Ruilope LM, Shennan A, Staessen JA, Tisler A, Waeber B, Zanchetti A, Mancia G; ESH Working Group on Blood Pressure Monitoring. European Society of Hypertension practice guidelines for home blood pressure monitoring. J Hum Hypertens. 2010 Dec;24(12):779-85. doi: 10.1038/jhh.2010.54. Epub 2010 Jun 3. PMID 20520631
- [Background] Komulainen S, Rintamaki H, Virokannas H, Keinanen-Kiukaanniemi S. Blood pressure responses to whole-body cold exposure: effect of metoprolol. J Hum Hypertens. 2004 Dec;18(12):905-6. doi: 10.1038/sj.jhh.1001758. No abstract available. PMID 15269706
- [Background] Bhaskaran K, Hajat S, Haines A, Herrett E, Wilkinson P, Smeeth L. Short term effects of temperature on risk of myocardial infarction in England and Wales: time series regression analysis of the Myocardial Ischaemia National Audit Project (MINAP) registry. BMJ. 2010 Aug 10;341:c3823. doi: 10.1136/bmj.c3823. PMID 20699305
- [Background] Sun Z. Cardiovascular responses to cold exposure. Front Biosci (Elite Ed). 2010 Jan 1;2(2):495-503. doi: 10.2741/e108. PMID 20036896
- [Background] Nayha S. Environmental temperature and mortality. Int J Circumpolar Health. 2005 Dec;64(5):451-8. doi: 10.3402/ijch.v64i5.18026. PMID 16440607
- [Result] Hintsala H, Kandelberg A, Herzig KH, Rintamaki H, Mantysaari M, Rantala A, Antikainen R, Keinanen-Kiukaanniemi S, Jaakkola JJ, Ikaheimo TM. Central aortic blood pressure of hypertensive men during short-term cold exposure. Am J Hypertens. 2014 May;27(5):656-64. doi: 10.1093/ajh/hpt136. Epub 2013 Aug 20. PMID 23964061
- [Derived] Hintsala HE, Kiviniemi AM, Antikainen R, Mantysaari M, Jokelainen J, Hassi J, Tulppo MP, Herzig KH, Keinanen-Kiukaanniemi S, Rintamaki H, Jaakkola JJK, Ikaheimo TM. High Home Blood Pressure Variability Associates With Exaggerated Blood Pressure Response to Cold Stress. Am J Hypertens. 2019 May 9;32(6):538-546. doi: 10.1093/ajh/hpz011. PMID 30984970
- [Derived] Hintsala H, Kentta TV, Tulppo M, Kiviniemi A, Huikuri HV, Mantysaari M, Keinanen-Kiukaannemi S, Bloigu R, Herzig KH, Antikainen R, Rintamaki H, Jaakkola JJ, Ikaheimo TM. Cardiac repolarization and autonomic regulation during short-term cold exposure in hypertensive men: an experimental study. PLoS One. 2014 Jul 1;9(7):e99973. doi: 10.1371/journal.pone.0099973. eCollection 2014. PMID 24983379